CLINICAL TRIAL: NCT06228963
Title: Orelabrutinib in the First-line Treatment of HP-positive Gastric MALT Lymphoma: a Multicenter, Open-label, Randomized Controlled Trial
Brief Title: Orelabrutinib in the Treatment of HP-positive Gastric MALT Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Yizhen Liu, Clinical Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: iNHL-02
Record Dates: First submitted 2024-01-12; First posted 2024-01-29 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: MALT Lymphoma of Stomach; Helicobacter Pylori Infection
MeSH Terms: interventions — orelabrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Triple therapy for eradication of Helicobacter Pylori+Orelabrutinib
  Interventions: Drug: Triple therapy for eradication of Helicobacter Pylori and Orelabrutinib
- Control group (Active Comparator): Triple therapy for eradication of Helicobacter Pylori
  Interventions: Drug: Triple therapy for eradication of Helicobacter Pylori

INTERVENTIONS:
Drug: Triple therapy for eradication of Helicobacter Pylori and Orelabrutinib — Triple therapy for H. pylori (oral administration for 2 weeks, followed by a 1-week break) plus Orelabrutinib for 8 weeks (or until progression, intolerable toxicity, death, or withdrawal from the study)
  Other Names: anti-HP and Orelabrutinib
  Arms: Experimental group
Drug: Triple therapy for eradication of Helicobacter Pylori — Triple therapy for H. pylori (oral administration for 2 weeks, followed by a 1-week break)
  Other Names: anti-HP
  Arms: Control group

SUMMARY:
Describe the efficacy and safety of Orelabrutinib in the treatment of HP-positive gastric MALT lymphoma

DETAILED DESCRIPTION:
This multicenter, open-label, randomized controlled trial is trying to evaluate the efficacy and safety of Orelabrutinib in the first-line treatment of HP-positive gastric MALT lymphoma

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Histologically confirmed gastric mucosa-associated lymphoid tissue (MALT) lymphoma;
* Current infection with Helicobacter pylori (Hp): Diagnosis can be made if any of the following criteria are met: a) Positive result in at least one of the following: RUT (rapid urease test), histological staining, or bacterial culture of gastric mucosal tissue; b) Positive result in 13C or 14C-UBT (urea breath test); c) Positive result in HpSA detection. A positive result in serum Hp antibody test indicates past infection, and patients who have never been treated can be considered as having current infection.
* ECOG (Eastern Cooperative Oncology Group) performance status 0-2.
* Lugano staging I-II1.
* Signed informed consent form.
* Evaluable lesions present.

Exclusion Criteria:

* Negative for Helicobacter pylori (HP);
* History of other tumors, except for cured cervical cancer or basal cell carcinoma of the skin;
* Patients with active HIV and syphilis infections;
* Pregnant or lactating women;
* Patients with severe active infections;
* Patients with multiple factors affecting oral medication (such as dysphagia, nausea, vomiting, chronic diarrhea, and intestinal obstruction);
* Other comorbidities or conditions that may prevent patients from completing the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
6-months CR rate | up to 6 months
  the ratio of numbers of patients with complete response to all the participants receiving treatment

SECONDARY OUTCOMES:
3-months CR rate | up to 3 months
  the ratio of numbers of patients with complete response to all the participants
2-year progression-free survival (PFS) | From date of patients sign informed consent until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
  the period from the date of patients sign informed consent to the observed progression of the disease or the occurrence of death for any reason
2-year event-free survival (EFS) | From date of patients sign informed consent until the date of first documented event, progression or date of death from any cause, whichever came first, assessed up to 2 years
  the period from the date of patients sign informed consent to the observed event for any reason
2-year overall survival rate | From date of patients sign informed consent until the date of death or the date of last follow-up time, whichever came first, assessed up to 2 years
  time between the date of patients sign informed consent and the date of death or the date of last follow-up time
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | Throughout the treatment period, up to 6 months
  Record the name of adverse events and number of participants with treatment-related adverse events as assessed by CTCAE v5.0

OTHER OUTCOMES:
Exploratory biomarkers | Throughout the treatment period, up to 2 years
  Biomarkers for predictive factors of efficacy at baseline or during the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Yizhen Liu, M.D., Ph.D., Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No